CLINICAL TRIAL: NCT06402396
Title: Assessing Pain by the painDETECT Questionnaire (PDQ) to Evaluate Drug Retention in Patients With Inflammatory Arthritis: A Danish Nationwide Prospective DANBIO Registry Study
Brief Title: Assessing Pain by the painDETECT Questionnaire (PDQ)
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Elisabeth Ginnerup-Nielsen, Post doctoral researcher, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: DANBIO PDQ
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Inflammatory Arthritis; Spondylarthropathies; Rheumatoid Arthritis; Psoriatic Arthritis
Keywords: Drug survival; Pain phenotypes; PainDETECT Questionnaire; Inflammatory Arthritis
MeSH Terms: conditions — Arthritis; Spondylarthropathies; Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-Neuropathic pain phenotype: Based on the PainDETECT Questionnaire (PDQ), patients scoring <13 will be classified as "exposed" as they are considered a group with non-neuropathic pain (Non-neuropathic pain phenotype)
  Interventions: Drug: bDMARDS
- Neuropathic pain phenotype: Based on the PainDETECT Questionnaire (PDQ), patients scoring ≥13 will be classified as "un-exposed" as they are considered a group with neuropathic pain (neuropathic pain phenotype)
  Interventions: Drug: bDMARDS

INTERVENTIONS:
Drug: bDMARDS — Patients at time of the PDQ assessment and up to 4 months thereafter being on ongoing bDMARDs treatment or on switch of bDMARD treatment.

SUMMARY:
Prospective cohort study using drug survival rates to assess the predictive value of the PDQ when used to classify patients into a non-neuropathic pain phenotype group (score <13) or a neuropathic pain phenotype group (score ≥13)

DETAILED DESCRIPTION:
The original painDETECT questionnaire (PDQ) DANBIO study was a survey among all DANBIO users having an arthritis diagnosis 'Pain and pain mechanisms in patients with inflammatory arthritis: A Danish nationwide cross-sectional DANBIO registry survey'. The PDQ was implemented onto the DANBIO touch screens for a period of 6 months in 2013-14 and data from more than 7000 individual patients were collected. The overall background for the study was that central pain mechanisms may be prominent in subsets of patients with rheumatoid arthritis (RA), psoriatic arthritis (PsA) and other spondyloarthritis (SpA). The study showed that approximately 50 % of patients experienced significant pain levels and that a high PDQ score was associated with higher levels of pain and DAS28 but not with markers of inflammatory activity such as CRP and swollen joint count. Furthermore, indications of more frequent bio-switch in the PDQ groups showing neuropathic pain features were found.

The aim of this study is to examine the association between drug retention of biological DMARDs (bDMARDs) and the PDQ pain classification categories (i.e. non-neuropathic vs. neuropathic features) and to investigate whether this categorization is predictive of drug retention and changes in clinical outcomes over a 5-year period.

ELIGIBILITY:
Inclusion Criteria:

* Registered in DANBIO
* Having inflammatory arthritis (Specific diagnoses include RA, PsA and other SpA)
* At time of the PDQ assessment and up to 4 months thereafter being on ongoing bDMARDs treatment or on switch of bDMARD treatment.

Exclusion Criteria:

- Missing answer to PDQ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients registered in DANBIO, having inflammatory arthritis (Specific diagnoses include RA, PsA and other SpA) and at time of the PDQ assessment and up to 4 months thereafter being on ongoing bDMARDs treatment or on switch of bDMARD treatment.
Sampling Method: Probability Sample
Enrollment: 7056 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Differences in bDMARDs drug retention rates | From baseline to 5 years followup
  Drug retention rates will be described using Kapan-Mayer curves. Differences in changes in bDMARDs drug retention rates over 5 years between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire.

SECONDARY OUTCOMES:
Differences in Patient acceptable symptom state (Pass) | From baseline to 5 years followup
  Differences in changes in patients having an acceptable symptom state at 5 years follow-up between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire.
  The PASS is defined as the highest symptom level below which a patient considers his/her symptom state as acceptable. it is answered via a yes or a no.
Differences in Swollen Joint Count (SJC, 0-28) | From baseline to 5 years followup
  Differences in changes in SJC 0-28 at 5 years follow-up between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire.
Differences in TenderJoint Count (TJC, 0-28) | From baseline to 5 years followup
  Differences in changes in TJC 0-28 at 5 years follow-up between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire.
Differences in Doctors' global assessment (VAS 0-100 mm.) | From baseline to 5 years followup
  Differences in changes in Doctors' global assessment 0-100 at 5 years follow-up between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire.
Differences in VAS pain (0-100 mm) (Higher indicates more pain) | From baseline to 5 years followup
  Differences in changes in VAS pain (0-100 mm) at 5 years follow-up between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire.
Differences in VAS fatigue (0-100 mm) (Higher indicates more fatigue) | From baseline to 5 years followup
  Differences in changes in VAS fatigue (0-100 mm) at 5 years follow-up between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire.
Differences in VAS global (0-100 mm) (Higher indicates more global disease activity) | From baseline to 5 years followup
  Differences in changes in VAS global (0-100 mm) at 5 years follow-up between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire.
Differences in HAQ (0-3) (higher indicates a more impaired functional level) | From baseline to 5 years followup
  Differences in changes in HAQ (0-3) at 5 years follow-up between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire. 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section the score given to that section is the worst score within the section, i.e. if one question is scored 1 and another 2, then the score for the section is 2. In addition, if an aide or device is used or if help is required from another individual, then the minimum score for that section is 2. If the section score is already 2 or more then no modification is made. The 8 scores of the 8 sections are summed and divided by 8. The result is the DI disability index index. In the event that one section is not completed by a subject then the summed score would be divided by 7.
Differences in CRP (mg/L) | From baseline to 5 years followup
  Differences in changes in CRP (mg/L) at 5 years follow-up between patients with a non-neuropathic phenotype and patients with a neuropathic pain phenotype based on the PainDETECT Questionnaire.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on RA diagnosis. | Measured at baseline
  The probability of having an RA diagnosis when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on PsA diagnosis. | Measured at baseline
  The probability of having an PsA diagnosis when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on SpA diagnosis. | Measured at baseline
  The probability of having an SpA diagnosis when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on number of bioswitches. | Measured at baseline
  The probability of having bioswitches when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on Swollen Joint Count (SJC, 0-28) | Measured at baseline
  The probability of having less swollen joints on the SJC 0-28 when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on TenderJoint Count (TJC, 0-28) | Measured at baseline
  The probability of having less tender joints on the TJC 0-28 when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on Doctors' global assessment (VAS: 0-100 mm) | Measured at baseline
  The probability of having a favourable score on Doctors' global assessment (VAS: 0-100 mm) when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on PASS (y/n) | Measured at baseline
  The probability of having an acceptable symptom state (PASS) when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on Patient acceptable symptom score (PASS (y/n)) | Measured at baseline
  The probability of having a favourable score on Patient acceptable symptom score (PASS) (yes/no) when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on VAS pain (0-100 mm) | Measured at baseline
  The probability of having a favourable score on VAS pain (0-100 mm) when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on VAS fatigue (0-100 mm) | Measured at baseline
  The probability of having a favourable score on VAS fatigue (0-100 mm) when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on VAS global (0-100 mm) | Measured at baseline
  The probability of having a favourable score on VAS global (0-100 mm) when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on the Health assessment questionnaire (HAQ (0-3)) | Measured at baseline
  The probability of having a favourable score on HAQ (0-3 mm) when having a non-neuropathic pain phenotype.
The prognostic value of pain phenotype classification by PainDETECT (PDQ) on C- reactive protein (CRP (mg/L)) | Measured at baseline
  The probability of having a favourable CRP when having a non-neuropathic pain phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine Amris, MD, DMSc, Study Chair — Bispebjerg and Frederiksberg Hospital

IPD SHARING:
Plan to Share IPD: No
Access to data can be granted upon reasonable request